CLINICAL TRIAL: NCT06744101
Title: Comparative Evaluation of Diffusion Weighted MRI And Ultrasonography In The Detection of Breast Lesions
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/013
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Breast LN

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Evaluate the effectiveness of Diffusion Weighted MRI (DWI) in detecting breast lesions. — Assess the sensitivity, specificity, and diagnostic accuracy of DWI compared to Ultrasonography (USG) for benign and malignant lesions.
Radiation: Compare Sensitivity and Specificity of DWI and USG — Analyze which modality performs better in lesion detection based on sensitivity and specificity.

SUMMARY:
This study aims to conduct a comparative evaluation of Diffusion Weighted MRI (DW-MRI) and Ultrasonography (US) in detecting breast lesions. Breast cancer remains a leading cause of cancer-related deaths among women worldwide, necessitating efficient and accurate diagnostic methods. Ultrasonography, a commonly used imaging modality, provides valuable insights into breast lesions but has limitations in sensitivity and specificity.

DETAILED DESCRIPTION:
Diffusion Weighted MRI, on the other hand, shows potential for higher accuracy in identifying malignant versus benign lesions due to its ability to assess tissue cellularity and integrity non-invasively. This research will involve a specified number of female participants within a defined age range, focusing on the comparative effectiveness, sensitivity, and specificity of DW-MRI and US. The findings are expected to contribute valuable insights into optimizing breast cancer diagnostic protocols, ultimately aiding in earlier detection, better patient outcomes, and possibly reducing the need for invasive biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women with suspected breast lesions
* Breast feeding woman
* Referred for MRI examination.
* Age 18 years or older
* Ability to provide informed consent.

Exclusion Criteria:

* Contraindications to MRI or contrast agent
* Previous breast Implant
* Early Pregnancy

Exclusion criteria

*

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Lesions
Study Population: Evaluation of Diffusion Weighted MRI And Ultrasonography In The Detection of Breast Lesions
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 12 Months
  * Ultrasonography (USG): BI-RADS classification.
  * Diffusion Weighted MRI (DWI): Apparent Diffusion Coefficient (ADC) values.
  * Scales/Measurements:
  * Sensitivity (%):
  Formula: (True Positives) ÷ (True Positives + False Negatives) × 100
  * Specificity (%):
  Formula: (True Negatives) ÷ (True Negatives + False Positives) × 100

CONTACTS AND LOCATIONS:
Locations (1):
- 563-B peoples colony 1 main satiana road Faisalabad, Faisalābad, Punjab Province, Pakistan